CLINICAL TRIAL: NCT02738411
Title: Influence of Intestinal Microbiota Implantation Parameters in the Neonatal Period in Premature Infants on Microbiota Profiles and Immune Orientation at 3 Years of Age
Brief Title: Influence of Intestinal Microbiota Implantation in Preterm Infants on Microbiota and Immune Orientation at 3 Years
Acronym: PrimiBiota
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: PHRC-I/2015/AF-01
Record Dates: First submitted 2016-04-11; First posted 2016-04-14 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Infant, Premature
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be drawn at 36 months for lymphocyte subpopulation characterization, stimulation tests and biobanking. Fecal samples at indicated time points will also be banked (bacterial rDNA will be extracted).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- The study population: The study population corresponds to infants born at less than 33 weeks of gestation.

SUMMARY:
The main objective of this research is to study the links between changes in the intestinal microbiota (in terms of diversity) during the first 6 weeks of life for preterm infants and the presence / absence of a TH1 immune status at 36 months of age.

DETAILED DESCRIPTION:
The secondary objectives are to study the links between changes of the intestinal microbiota premature infants in terms of:

* changing diversity of the microbiota in the first 6 weeks of life;
* changes in the bacterial community (UniFrac study) during the first 6 weeks of life;
* diversity of the microbiota up to 6 weeks;

-AND-

* diversity of the microbiota at 1, 2 & 3 years;
* bacterial communities (UniFrac study) at 1, 2 & 3 years;
* lymphocyte subpopulation profiles at 3 years;
* serum immunoglobulin A, G, M, E levels at 3 years;
* history of infectious episodes, allergic and inflammatory episodes during the first 3 years of life.

The links between certain variables known in the literature and neonatal microbiota will be confirmed / studied in our population:

* mode of delivery;
* length (and type) of antibiotic therapy in the neonatal period;
* duration of breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* The parents of the patient (or legal guardian if any) have been informed about the implementation of the study, its objectives, its constraints, and patient rights
* The parents of the patient (or legal guardian if any) must have given their free and informed consent and signed the consent form
* The patient must be affiliated with or beneficiary of a health insurance plan
* Premature infants born at less than 33 weeks of gestation

Exclusion Criteria:

* The patient is participating in another interventional study (Excepted " Recherche du Portage de Clostridium butyricum et de Toxines de Clostridium chez les Prématurés Hospitalisés en Néonatologie afin de prédire la survenue d'Entérocolites Nécrosantes", RCB 2016-A00-529-42 ; " BetaDose Dose reduction of antenatal betamethasone given to prevent the neonatal complications associated with very preterm birth ", RCB 2016-001486-90.
* It is not possible to correctly inform the parent (or legal guardian, if applicable)
* A serious deformity or digestive malformation was diagnosed at birth
* During the hospital stay in the neonatology department, the patient had a digestive disease requiring surgery (except necrotizing enterocolitis)
* A transfer to another hospital is foreseen/predictable (eg, due to geographical distance)

Max Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population consists of premature babies born at < 33 months gestation.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The presence/absence of a Th1 type immune orientation | 36 months
  Immune orientation will be determined according to the following ratio determined by lymphocyte stimulation tests: INF-gamma/(INF-gamma+IL+4). The latter ratio varies between 0 and 0.5 with IL-4 > INF-gamma (TH2 orientation) and between 0.5 and 1 when INF-gamma > IL-4 (TH1 orientation).

SECONDARY OUTCOMES:
Blood lymphocyte subset determination | 36 months
  Subsets are determined according to the presence/absence of the following differentiation clusters: CD3, CD4, CD8, CD19, CD25, CD56, CD127, FOXP3.

OTHER OUTCOMES:
Serum Immunoglobulin A level | 36 months
Serum Immunoglobulin G level | 36 months
Serum Immunoglobulin M level | 36 months
Serum Immunoglobulin E level | 36 months
The number of days in good health and no medications | 36 months
Richness of fecal microbiota (number of operational taxonomic units observed) | Day 0 (first meconium)
Richness of fecal microbiota (number of operational taxonomic units observed) | Week 1
Richness of fecal microbiota (number of operational taxonomic units observed) | Week 2
Richness of fecal microbiota (number of operational taxonomic units observed) | Week 3
Richness of fecal microbiota (number of operational taxonomic units observed) | Week 4
Richness of fecal microbiota (number of operational taxonomic units observed) | Week 5
Richness of fecal microbiota (number of operational taxonomic units observed) | Week 6
Richness of fecal microbiota (number of operational taxonomic units observed) | 12 months
Richness of fecal microbiota (number of operational taxonomic units observed) | 24 months
Richness of fecal microbiota (number of operational taxonomic units observed) | 36 months
Diversity of fecal microbiota (Shannon's index) | Day 0 (first meconium)
Diversity of fecal microbiota (Shannon's index) | Week 1
Diversity of fecal microbiota (Shannon's index) | Week 2
Diversity of fecal microbiota (Shannon's index) | Week 3
Diversity of fecal microbiota (Shannon's index) | Week 4
Diversity of fecal microbiota (Shannon's index) | Week 5
Diversity of fecal microbiota (Shannon's index) | Week 6
Diversity of fecal microbiota (Shannon's index) | 12 months
Diversity of fecal microbiota (Shannon's index) | 24 months
Diversity of fecal microbiota (Shannon's index) | 36 months
Functional richness of fecal microbiota (number of functional groups observed) | Day 0 (first meconium)
  Functional groups are determined via the classification of each OTU according to the following factors: 1) pathogenicity (pathogen/intermediate/commensal); 2) aerobic versus anaerobic; 3) Cocci + versus others.
Functional richness of fecal microbiota (number of functional groups observed) | Week 1
  Functional groups are determined via the classification of each OTU according to the following factors: 1) pathogenicity (pathogen/intermediate/commensal); 2) aerobic versus anaerobic; 3) Cocci + versus others.
Functional richness of fecal microbiota (number of functional groups observed) | Week 2
  Functional groups are determined via the classification of each OTU according to the following factors: 1) pathogenicity (pathogen/intermediate/commensal); 2) aerobic versus anaerobic; 3) Cocci + versus others.
Functional richness of fecal microbiota (number of functional groups observed) | Week 3
  Functional groups are determined via the classification of each OTU according to the following factors: 1) pathogenicity (pathogen/intermediate/commensal); 2) aerobic versus anaerobic; 3) Cocci + versus others.
Functional richness of fecal microbiota (number of functional groups observed) | Week 4
  Functional groups are determined via the classification of each OTU according to the following factors: 1) pathogenicity (pathogen/intermediate/commensal); 2) aerobic versus anaerobic; 3) Cocci + versus others.
Functional richness of fecal microbiota (number of functional groups observed) | Week 5
  Functional groups are determined via the classification of each OTU according to the following factors: 1) pathogenicity (pathogen/intermediate/commensal); 2) aerobic versus anaerobic; 3) Cocci + versus others.
Functional richness of fecal microbiota (number of functional groups observed) | Week 6
  Functional groups are determined via the classification of each OTU according to the following factors: 1) pathogenicity (pathogen/intermediate/commensal); 2) aerobic versus anaerobic; 3) Cocci + versus others.
Functional richness of fecal microbiota (number of functional groups observed) | 12 months
  Functional groups are determined via the classification of each OTU according to the following factors: 1) pathogenicity (pathogen/intermediate/commensal); 2) aerobic versus anaerobic; 3) Cocci + versus others.
Functional richness of fecal microbiota (number of functional groups observed) | 24 months
  Functional groups are determined via the classification of each OTU according to the following factors: 1) pathogenicity (pathogen/intermediate/commensal); 2) aerobic versus anaerobic; 3) Cocci + versus others.
Functional richness of fecal microbiota (number of functional groups observed) | 36 months
  Functional groups are determined via the classification of each OTU according to the following factors: 1) pathogenicity (pathogen/intermediate/commensal); 2) aerobic versus anaerobic; 3) Cocci + versus others.
Functional diversity of fecal microbiota (Shannon's index) | Day 0 (first meconium)
  Functional groups are determined via the classification of each OTU according to the following factors: 1) pathogenicity (pathogen/intermediate/commensal); 2) aerobic versus anaerobic; 3) Cocci + versus others.
Functional diversity of fecal microbiota (Shannon's index) | Week 1
  Functional groups are determined via the classification of each OTU according to the following factors: 1) pathogenicity (pathogen/intermediate/commensal); 2) aerobic versus anaerobic; 3) Cocci + versus others.
Functional diversity of fecal microbiota (Shannon's index) | Week 2
  Functional groups are determined via the classification of each OTU according to the following factors: 1) pathogenicity (pathogen/intermediate/commensal); 2) aerobic versus anaerobic; 3) Cocci + versus others.
Functional diversity of fecal microbiota (Shannon's index) | Week 3
  Functional groups are determined via the classification of each OTU according to the following factors: 1) pathogenicity (pathogen/intermediate/commensal); 2) aerobic versus anaerobic; 3) Cocci + versus others.
Functional diversity of fecal microbiota (Shannon's index) | Week 4
  Functional groups are determined via the classification of each OTU according to the following factors: 1) pathogenicity (pathogen/intermediate/commensal); 2) aerobic versus anaerobic; 3) Cocci + versus others.
Functional diversity of fecal microbiota (Shannon's index) | Week 5
  Functional groups are determined via the classification of each OTU according to the following factors: 1) pathogenicity (pathogen/intermediate/commensal); 2) aerobic versus anaerobic; 3) Cocci + versus others.
Functional diversity of fecal microbiota (Shannon's index) | Week 6
  Functional groups are determined via the classification of each OTU according to the following factors: 1) pathogenicity (pathogen/intermediate/commensal); 2) aerobic versus anaerobic; 3) Cocci + versus others.
Functional diversity of fecal microbiota (Shannon's index) | 12 months
  Functional groups are determined via the classification of each OTU according to the following factors: 1) pathogenicity (pathogen/intermediate/commensal); 2) aerobic versus anaerobic; 3) Cocci + versus others.
Functional diversity of fecal microbiota (Shannon's index) | 24 months
  Functional groups are determined via the classification of each OTU according to the following factors: 1) pathogenicity (pathogen/intermediate/commensal); 2) aerobic versus anaerobic; 3) Cocci + versus others.
Functional diversity of fecal microbiota (Shannon's index) | 36 months
  Functional groups are determined via the classification of each OTU according to the following factors: 1) pathogenicity (pathogen/intermediate/commensal); 2) aerobic versus anaerobic; 3) Cocci + versus others.
The relative abundance of primary fecal microbiota families | Day 0 (first meconium)
The relative abundance of primary fecal microbiota families | Week 1
The relative abundance of primary fecal microbiota families | Week 2
The relative abundance of primary fecal microbiota families | Week 3
The relative abundance of primary fecal microbiota families | Week 4
The relative abundance of primary fecal microbiota families | Week 5
The relative abundance of primary fecal microbiota families | Week 6
The relative abundance of primary fecal microbiota families | 12 months
The relative abundance of primary fecal microbiota families | 24 months
The relative abundance of primary fecal microbiota families | 36 months
Fecal microbiota unifrac ordination score | Day 0 (first meconium)
Fecal microbiota unifrac ordination score | Week 1
Fecal microbiota unifrac ordination score | Week 2
Fecal microbiota unifrac ordination score | Week 3
Fecal microbiota unifrac ordination score | Week 4
Fecal microbiota unifrac ordination score | Week 5
Fecal microbiota unifrac ordination score | Week 6
Fecal microbiota unifrac ordination score | 12 months
Fecal microbiota unifrac ordination score | 24 months
Fecal microbiota unifrac ordination score | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne Filleron, MD, PhD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (3):
- France (3):
  - CHRU de Montpellier - Hôpital Arnaud de Villeneuve, Montpellier
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - Réseau GRANDIR EN LANGUEDOC-ROUSILLON, Saint-Gély-du-Fesc